CLINICAL TRIAL: NCT00039975
Title: Evaluation of Potential Pharmacokinetic Interactions Between HIV Protease Inhibitors and Calcium Channel Blockers
Brief Title: Interactions Between HIV Protease Inhibitors and Calcium Channel Blockers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A5159; 10959 (Registry Identifier: DAIDS ES); ACTG A5159; AACTG A5159
Record Dates: First submitted 2002-06-18; First posted 2002-06-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Cardiovascular Diseases; Hypertension
Keywords: Drug Interactions; HIV Protease Inhibitors; Ritonavir; Indinavir; Calcium Channel Blockers; Pharmacokinetics; Diltiazem; Amlodipine
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Hypertension | interventions — Indinavir; Ritonavir; Amlodipine; Diltiazem

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Amlodipine
Drug: Diltiazem HCl

SUMMARY:
Diltiazem CD and amlodipine are drugs used to treat heart disease and high blood pressure. The purpose of this study is to find out if these drugs interact with the anti-HIV drugs indinavir and ritonavir. The study will also look at the safety of taking the study drugs together.

Heart disease and high blood pressure are major health concerns for people with HIV. Standard treatment for these illnesses often includes calcium channel blockers (CCBs). There is a potential for significant drug interactions between CCBs and HIV protease inhibitors (PIs) that may influence the dosing, monitoring, and choosing of CCBs and PIs when used in people infected with HIV. This study will examine the drug interactions between 2 commonly used CCBs and the PI combination indinavir and ritonavir (IDV/RTV). This information should help doctors choose the appropriate treatment for high blood pressure or heart disease in people taking PIs.

DETAILED DESCRIPTION:
Ischemic cardiovascular disease and hypertension occur in persons with HIV infection, and the incidence and prevalence may increase over time as the infected population ages. Standard pharmacologic interventions for these illnesses often include calcium channel blockers (CCBs). Many of the calcium channel blockers are metabolized by cytochrome P450 3A4 (CYP 3A4), which is inhibited by some protease inhibitors (PIs). Thus, there is potential for clinically significant interactions between CCBs and PIs. The presence of significant drug-drug interactions may influence the dosing, monitoring, and choosing of CCBs and/or PIs when used in persons with HIV infection. Because of the potential concomitant use of CCBs with the PI combination IDV/RTV, this study will evaluate bi-directional drug-drug interactions between 2 commonly used CCBs and IDV/RTV. This information should assist clinicians in choosing the appropriate CCBs to treat hypertension or cardiovascular disease in persons taking PIs.

Patients are randomized to 1 of the following 2 arms:

Arm A: diltiazem CD interaction with IDV and RTV. Arm B: amlodipine interaction with IDV and RTV. From Days 1 to 7, patients take diltiazem CD (Arm A) or amlodipine (Arm B). Plasma is collected for PK over a 24-hour period beginning on Day 7. From Days 8 to 19, patients stop taking their assigned CCB and take IDV and RTV. Plasma is collected for PK over a 12-hour period on Day 19. From Days 20 to 26, patients continue to take IDV and RTV and add diltiazem CD (Arm A) or amlodipine (Arm B). Patients stop all 3 drugs after the last dose on Day 26. Plasma is collected for PK for a 24-hour period beginning on Day 26. Blood work, liver and kidney function tests, urinalysis, and an electrocardiogram (EKG) are performed at some visits.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-negative.
* Are between the ages of 18 and 60.
* Agree not to become pregnant or to impregnate and to use an acceptable form of contraception while receiving study drugs and for 1 month after stopping study drugs. Patients who are not of reproductive potential are eligible without the contraception requirement.
* Are within 30 percent of ideal body weight.
* Weigh at least 110 lbs.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have a history of any illness that requires current medical therapy.
* Have a history of any kidney disorder.
* Have any medical condition that, in the opinion of the investigator, would interfere with the study.
* Are pregnant or breast-feeding.
* Use certain drugs within 14 days prior to study entry.
* Are allergic or sensitive to study drugs.
* Use drugs or alcohol in a way which, in the opinion of the investigator, would interfere with the study.
* Have any abnormality on electrocardiogram within 21 days prior to study entry.
* Participate in any investigational drug studies within 21 days prior to study entry and during study.
* Are unable to participate in pharmacokinetic visits.
* Are unable to understand or follow the fluid intake requirement during the periods of IDV/RTV administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Glesby, Study Chair
Locations (9):
- United States (9):
  - Univ of California San Francisco, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ (St. Louis), St Louis, Missouri
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Background] Yunis NA, Stone VE. Cardiac manifestations of HIV/AIDS: a review of disease spectrum and clinical management. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Jun 1;18(2):145-54. doi: 10.1097/00042560-199806010-00006. PMID 9637579
- [Background] Henry K, Melroe H, Huebsch J, Hermundson J, Levine C, Swensen L, Daley J. Severe premature coronary artery disease with protease inhibitors. Lancet. 1998 May 2;351(9112):1328. doi: 10.1016/S0140-6736(05)79053-X. No abstract available. PMID 9643798
- [Background] Cattelan AM, Trevenzoli M, Sasset L, Rinaldi L, Balasso V, Cadrobbi P. Indinavir and systemic hypertension. AIDS. 2001 Apr 13;15(6):805-7. doi: 10.1097/00002030-200104130-00021. No abstract available. PMID 11371700
- [Background] Passalaris JD, Sepkowitz KA, Glesby MJ. Coronary artery disease and human immunodeficiency virus infection. Clin Infect Dis. 2000 Sep;31(3):787-97. doi: 10.1086/313995. Epub 2000 Oct 4. PMID 11017831
- [Result] Glesby MJ, Aberg JA, Kendall MA, Fichtenbaum CJ, Hafner R, Hall S, Grosskopf N, Zolopa AR, Gerber JG; Adult AIDS Clinical Trials Group A5159 Protocol Team. Pharmacokinetic interactions between indinavir plus ritonavir and calcium channel blockers. Clin Pharmacol Ther. 2005 Aug;78(2):143-53. doi: 10.1016/j.clpt.2005.04.005. PMID 16084849